CLINICAL TRIAL: NCT02474108
Title: Pilot, Randomized,Single Blind Trial of Surgical Prevention of Atrial Fibrillation in Patients With Rheumatic Mitral Valve Lesion
Brief Title: Surgical Prevention of Atrial Fibrillation in Patients With Rheumatic Mitral Valve Lesion and Left Atrium Enlargement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: SPAF
Record Dates: First submitted 2015-04-23; First posted 2015-06-17 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation; Rheumatic Heart Disease
Keywords: atrial fibrillation; radiofrequency ablation; prevention of AF; mitral valve; left atrium enlargement; cryoablation
MeSH Terms: conditions — Atrial Fibrillation; Rheumatic Heart Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without prevention (Placebo Comparator): isolated mitral valve replacement or reconstruction, implantation of cardiac monitor
  Interventions: Device: cardiomonitor
- group of prevention (Active Comparator): mitral valve replacement or reconstruction with surgical prevention of AF (concomitant ablation of the left atrium) and implantation of cardiac monitor.
  Prophylactic surgical ablation is performed to prevent AF in patients during mitral valve surgery. Ablation is performed by radiofrequency electrode or cryoprobe.
  Interventions: Procedure: surgical prevention of atrial fibrillation; Device: cardiomonitor

INTERVENTIONS:
Procedure: surgical prevention of atrial fibrillation — Prophylactic surgical ablation is performed to prevent AF in patients during mitral valve surgery. Ablation is performed by radiofrequency electrode or cryoprobe. Pulmonary veins, posterior wall of the left atrium will be isolated by the scheme box-lesion with additional lines to the mitral valve and appendage of left atrium.
  Arms: group of prevention
Device: cardiomonitor — in both groups cardiac rhythm will be controlled by a cardiomonitor

SUMMARY:
This study evaluates the safety and efficiency of surgical prevention of atrial fibrillation in patients with valvular heart disease and left atrium enlargement

DETAILED DESCRIPTION:
Preservation or appearance of AF(atrial fibrillation) after mitral valve surgery substantially reduce the number of excellent and good results of the operation in the long-term period, causing circulatory insufficiency, increased pulmonary hypertension, increasing the risk of thromboembolic events and stroke.

Significant predictors of AF after surgery are the initial size of the left atrium more than 6.0 cm, stenotic lesions and rheumatic genesis of mitral defect. 80% of patients in this group had AF during the first year after operation.

ELIGIBILITY:
Inclusion Criteria:

* rheumatic mitral valve lesion
* the absence a history of AF
* sinus rhythm
* left atrium size more than 6.0 cm

Exclusion Criteria:

* refusal to participate in the study
* aortic stenosis / regurgitation
* coronary atherosclerosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
composite outcome measure of complications | up to 1 year

SECONDARY OUTCOMES:
number of participants with freedom from AF according to the long-term ECG monitoring | 1 year
transport function of the left atrium according to TTE (transthoracic echo) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- MeshalkinRI, Novosibirsk, Russia